CLINICAL TRIAL: NCT00179530
Title: The Effect of Relaxation Response Training on Declarative Memory and Salivary Cortisol in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2001-P-002249
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Behavioral: Relaxation Response — Relaxation training

SUMMARY:
To evaluate whether a 5-week relaxation response intervention influences the learning, memory or attention of healthy older adults.

ELIGIBILITY:
Inclusion Criteria:

* 65 to 80 years od age
* No prior or current psychiatric or neurological condition.
* score above 24 on the Mini-Mental State Exam (MMSE)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 1999-05; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Evaluate whether a RR training program would decrease anxiety levels, improve attention, declarative memory performance in healthy older adults. | 8 weeks

SECONDARY OUTCOMES:
Evaluate whether a RR training program would decrease salivary cortisol levels in healthy older adults. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery A Dusek, PhD, Principal Investigator — Beth Israel Deaconess Medical Center, Mind/Body Medical Institute